CLINICAL TRIAL: NCT01248013
Title: Outcome Effectiveness Predictors of Irritable Bowel Syndrome Hypnotherapy
Brief Title: Irritable Bowel Syndrome Hypnotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mind-Body Digestive Center (Other)
Responsible Party: Charles D. Gerson, M.D., Mind-Body Digestive Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0575
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Results first posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: gut focused hypnotherapy — 7 session hypnotherapy protocol designed for irritable bowel syndrome

SUMMARY:
The primary goal of the study was whether gut focused hypnotherapy, in a group format, was successful in reduction of symptoms in patients with irritable bowel syndrome. The secondary goal was to see if any outcome predictors could be determined.

DETAILED DESCRIPTION:
Patients with Irritable Bowel Syndrome entering a group hypnotherapy program are asked to complete a series of questionnaires at the outset, and repeat a symptom severity scale at intervals over the one year period after termination of treatment. Eligibility was limited to patients with age greater than 20.

Outcome measures were improvement in symptom score. Outcome predictors studied included quality of relationships, measured with a Quality of Relationship Inventory and attribution of IBS to physical or emotional cause, measured with a Mind-Body IBS Questionnaire, both administered before onset of hypnotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of irritable bowel syndrome by Rome II criteria, age 20 and older

Exclusion Criteria:

* Age below 20

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mind Body Digestive Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at their initial visit to an IBS treatment center, on a purely voluntary basis into a group hypnotherapy program, from 2005 to 2009. 75 patients were entered into the study. Another 14 filled out initial questionnaires but then declined to enter treatment or dropped out after 1 or 2 sessions.
Pre-assignment Details: There was no control group assignment in this preliminary study which was designed to see if hypnotherapy, already proven effective in individual treatment was effective when using a group format.
Groups:
- Group Hypnotherapy for Irritable Bowel Syndrome: IBS subjects, in groups of 3 to 8 participants, received a specific gut focused hypnotherapy protocol. Meetings were bi-weekly, seven in all, and each meeting was 45 minutes in length. CD's were distributed for use at home between meetings.
Period: Overall Study
Arm/Group | Group Hypnotherapy for Irritable Bowel Syndrome
Started | 89
Irritable Bowel Syndrome Hypnotherapy | 75
Completed | 75
Not Completed | 14
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Arm/Group | Group Hypnotherapy for Irritable Bowel Syndrome
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 89

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Group Hypnotherapy in Irritable Bowel Syndrome
Description: assessed by symptom severity scale given before treatment began and after 7 bi-weekly sessions, at 3 months, 6 months and 12 months
Time Frame: one year
Reporting Status: Not Posted

2. Secondary Outcome: Outcome Predictors
Description: to determine whether relationship quality, or attribution of symptoms to physical or emotional causation correlated with result
Time Frame: one year
Reporting Status: Not Posted

3. Primary Outcome: Percentage of Patients With Significant Reduction in Their IBS Symptom Severity Score One Year After Completion of Therapy.
Description: The IBS Symptom Severity Scale has four components, severity of abdominal pain, number of days with pain in past 10 days, abdominal distension, bowel habit and interference with life in general. Maximum score is 500, minimum score is 0. The lower the score, the lower the symptom severity. Participants are considered clinically improved if they have a reduction in score of 50 points or greater.
Time Frame: One year after termination of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Group Hypnotherapy for Irritable Bowel Syndrome
Number analyzed (Participants) | 89
percentage of participants | 60

ADVERSE EVENTS:
Arm/Group | Group Hypnotherapy for Irritable Bowel Syndrome
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 0/89

LIMITATIONS AND CAVEATS:
Subjects who dropped out did so for reasons of inconvenience of scheduling attendance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No